CLINICAL TRIAL: NCT02495285
Title: Infusion of Gelatine Solutions in Pediatric Patients Aged up to 12 Years
Brief Title: Gelatines in Pediatric PatientS
Acronym: GPS
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-1406
Record Dates: First submitted 2015-06-12; First posted 2015-07-13 (Estimated); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Treatment of Hypovolemia and Shock
Keywords: pediatric patients gelatine
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gelofusine 4%: Children age ≤ 12 years
  Interventions: Drug: Gelofusine 4%
- Gelaspan 4%: Children age ≤ 12 years
  Interventions: Drug: Gelaspan 4%

INTERVENTIONS:
Drug: Gelofusine 4%
  Groups: Gelofusine 4%
Drug: Gelaspan 4%
  Groups: Gelaspan 4%

SUMMARY:
The aim of volume replacement is to compensate a reduction in the intravascular volume e.g. during surgery and to counteract hypovolemia in order to maintain hemodynamics and vital functions. So far, there is only few data on the safety and efficacy of the products under investigation in children.

The primary aim of this non-interventional observational study (NIS) is to collect further data of gelatine solutions in a large pediatric population during routine clinical practice.

ELIGIBILITY:
Inclusion:

* Age ≤ 12 years
* American Society of Anesthesiologists (ASA) risk score: ≤ III
* Peri-operative infusion of gelatine solutions
* Informed consent and/or data protection declaration signed by parents/legal guardians (according to local requirements)

Exclusion:

* Inclusion in another investigational study in the field of volume replacement which could interfere with the routine clinical practice regarding the administration of the gelatine solutions
* In addition contraindications as outlined in the valid local Summaries of Product Characteristics (SmPCs) have to be considered.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2015-05; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sümpelmann, Prof., Principal Investigator — Medizinische Hochschule Hannover (MHH)
Locations (11):
- National Cardiology Hospital, Sofia, Bulgaria
- Germany (4):
  - Auf der Bult, Hanover
  - Medizinische Hochschule Hannover, Pädiatrische Kardiologie und Intensivmedizin, Hanover
  - Klinik Hallerwiese/Cnopf´sche Kinderklinik, Nuremberg
  - Klinikum Stuttgart, Olgahospital und Frauenklinik, Stuttgart
- Italy (2):
  - Azienda Policlinico Universitaria G. Rodolico -Vittorio Emanuele, Catania
  - Ospedale dei Bambini Vittore Buzzi, Milan
- Spain (3):
  - Hospital de Sant Joan de Déu, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Son Espases, Palma de Mallorca
- Alder Hey Children's NHS FT, Liverpool, United Kingdom

REFERENCES:
- [Derived] Rudolf D, Witt L, Boethig D, Rigterink V, Zander R, Sumpelmann R, Dennhardt N. The impact of modified fluid gelatin 4% in a balanced electrolyte solution on plasma osmolality in children-A noninterventional observational study. Paediatr Anaesth. 2022 Aug;32(8):961-966. doi: 10.1111/pan.14494. Epub 2022 May 31. PMID 35588274

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolment target of 1500 patients was not met due to slow recruitment although duration of study had been extended to 60 months
Groups:
- Gelofusine 4%: Children age ≤ 12 years
  Gelofusine 4%
- Gelaspan 4%: Children age ≤ 12 years
  Gelaspan 4%
Period: Overall Study
Arm/Group | Gelofusine 4% | Gelaspan 4%
Started | 121 | 480
Completed | 121 | 480
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gelofusine 4% | Gelaspan 4% | Total
Number analyzed (Participants) | 121 | 480 | 601
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 121 | 480 | 601
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 52.6 (45.70) | 23.15 (34.12) | 29.08 (38.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 203 | 249
  Male | 75 | 277 | 352
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 53 | 6 | 59
  United Kingdom | 8 | 0 | 8
  Bulgaria | 30 | 0 | 30
  Germany | 20 | 431 | 451
  Spain | 10 | 43 | 53

OUTCOME MEASURES:

1. Primary Outcome: Dosing of the Products During Surgery
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
ml/kg | 14.58 (6.85) | 12.64 (4.72)

2. Secondary Outcome: Potentia Hydrogenii
Description: Potentia hydrogenii (ph) was part of blood sampling/laboratory to measure the levels of oxygen and carbon dioxide.
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for potentia hydrogenii were not entered for all partipants by the sites in the data collection form.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
unitless
  Before Infusion: number analyzed (Participants) | 107 | 438
  Before Infusion | 7.35 (0.08) | 7.34 (0.06)
  After Infusion: number analyzed (Participants) | 110 | 447
  After Infusion | 7.34 (0.07) | 7.32 (0.07)

3. Secondary Outcome: Hemoglobin
Description: mmol/L
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for Hemoglobin were not entered for all participants by the sites in the data collection form.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
mmol/L
  Before Infusion: number analyzed (Participants) | 90 | 441
  Before Infusion | 11.02 (2.51) | 11.35 (2.22)
  After infusion: number analyzed (Participants) | 93 | 448
  After infusion | 10.01 (2.42) | 10.30 (2.16)

4. Secondary Outcome: Lactate
Description: mmol/l
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for lactates were not entered for all participants by the sites in the data collection form.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
mmol/l
  Before infusion: number analyzed (Participants) | 106 | 430
  Before infusion | 1.38 (0.80) | 1.19 (0.62)
  After infusion: number analyzed (Participants) | 108 | 440
  After infusion | 1.48 (0.87) | 1.30 (0.82)

5. Secondary Outcome: Hematocrit
Description: %
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for Hematocrit were not entered for all subjects by the sites in the data collection form.
Measure: Mean (Standard Error); unit: "%"
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
"%"
  Before infusion: number analyzed (Participants) | 68 | 425
  Before infusion | 35.33 (6.76) | 35.06 (6.92)
  After infusion: number analyzed (Participants) | 71 | 433
  After infusion | 31.67 (7.64) | 32.07 (7.12)

6. Secondary Outcome: Glucose
Description: mmol/l
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for glucose were not entered for all participants by the sites in the data collection form
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
mmol/l
  Before infusion: number analyzed (Participants) | 106 | 434
  Before infusion | 6.13 (3.02) | 5.21 (1.18)
  After infusion: number analyzed (Participants) | 109 | 441
  After infusion | 6.83 (4.36) | 6.61 (1.96)

7. Secondary Outcome: Serum Prolin
Description: µmol/l
Time Frame: Before (0 - 2 days) and up to 2 days after infusion of gelatin solutions
Population: Serum proline was only documented in four study participants in total. Not part of clinical routine.
Measure: Mean (Standard Deviation); unit: µmol/l
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
µmol/l
  Before infusion: number analyzed (Participants) | 4 | 0
  Before infusion | 235.25 (2.5) |
  After infusion: number analyzed (Participants) | 4 | 0
  After infusion | 180 (43.63) |

8. Secondary Outcome: Serum Creatinine
Description: µmol/l
Time Frame: Before (0 - 2 days) and up to 2 days after infusion of gelatin solutions
Population: The data for Serum Creatinine were not entered for all participants by the sites in the data collection form.
Measure: Mean (Standard Deviation); unit: µmol/l
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
µmol/l
  Before infusion: number analyzed (Participants) | 92 | 387
  Before infusion | 30.92 (15.32) | 31.08 (16.48)
  After infusion: number analyzed (Participants) | 87 | 318
  After infusion | 30.23 (14.06) | 33.13 (17.80)

9. Secondary Outcome: Number of Participants With (Serious) Adverse Events / Reactions
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Measure: Count of Participants; unit: Participants
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
Participants | 1 | 4

10. Secondary Outcome: Heart Rate
Description: beats per minute
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for heart rate were not entered for all participants by the sites in the data collection form.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
beats per minute
  Before infusion: number analyzed (Participants) | 120 | 480
  Before infusion | 116.74 (25.72) | 121.20 (22.54)
  After infusion: number analyzed (Participants) | 119 | 479
  After infusion | 113.24 (22.54) | 118.72 (21.88)

11. Secondary Outcome: Mean Arterial Pressure
Description: mmHg
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Population: The data for mean arterial pressure were not entered for all participants by the sites in the data collection form
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
mmHg
  Before infusion: number analyzed (Participants) | 120 | 478
  Before infusion | 58.03 (14.81) | 46.72 (11.54)
  After infusion: number analyzed (Participants) | 119 | 478
  After infusion | 65.23 (14.48) | 55.55 (11.25)

12. Secondary Outcome: Follow-up Assessed by Number of Participants With Post-operative Complications
Time Frame: At discharge from the hospital or in-hospital 3 months after start of gelatine infusion, whatever occurs first.
Measure: Count of Participants; unit: Participants
Arm/Group | Gelofusine 4% | Gelaspan 4%
Number analyzed (Participants) | 121 | 480
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Before (0 - 2 h) and up to 2 h after infusion of gelatin solutions
Arm/Group | Gelofusine 4% | Gelaspan 4%
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/480
Serious Adverse Events (participants affected / at risk) | 0/121 | 1/480
Other Adverse Events (participants affected / at risk) | 1/121 | 3/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelofusine 4% (N=121) | Gelaspan 4% (N=480)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gelofusine 4% (N=121) | Gelaspan 4% (N=480)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Electrolyte imblance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemodilution (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02495285/Prot_SAP_000.pdf